CLINICAL TRIAL: NCT06828211
Title: Prospective Open Randomized Controlled Trial on the Effectiveness and Tolerability of Trans-resveratrol (derived from Polygonum Cuspidatum Root Extr.) on the Development of CHF in Postmenopausal Women with HTN and Reduced BMD
Brief Title: Trans-resveratrol's Influence on the Development of CHF in Early Postmenopausal Women with HTN and Reduced BMD
Acronym: Not aplicable
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OMNIFARMA LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27/08-1/OD/PD; Was not given (Other: Omnifarma LLC)
Record Dates: First submitted 2025-01-15; First posted 2025-02-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Arterial Hypertension; Osteopenia; Menopause
MeSH Terms: conditions — Heart Failure; Hypertension; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group recieving the intervention as Trans-resveratrol extract from Polygonum Cuspidatum (Active Comparator): Study group recieving the intervention as Trans-resveratrol extract from Polygonum Cuspidatum has been assigned Trans-resveratrol extract from Polygonum Cuspidatum intervention - 50 patients, female postmenopausal (1-4 years) with hypertension (stage I-II) and decreased bone mineral density
  Interventions: Dietary Supplement: Trans-resveratrol extract from Polygonum Cuspidatum
- Placebo group (Placebo Comparator): Placebo group - 30 patients, female postmenopausal (1-4 years) with hypertension (stage I-II) and decreased bone mineral density
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Trans-resveratrol extract from Polygonum Cuspidatum — Trans-resveratrol extract from Polygonum Cuspidatum
  Arms: Study group recieving the intervention as Trans-resveratrol extract from Polygonum Cuspidatum
Other: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
1. To measure the ability of trans-resveratrol to influence the development of chronic heart failure (CHF) in women in the early postmenopausal period (1-4 years) with hypertension (HTN) and reduced bone mineral density (BMD).
2. To evaluate the safety of long-term use of trans-resveratrol in an amount of 500 mg per day.
3. To develop modern measures to influence the development of CHF in women of this group

ELIGIBILITY:
Inclusion Criteria:

* availability of a signed Informed Consent (Information Sheet) of the patient to participate in the clinical trial;
* female patients in the postmenopausal period (1-4 years) with hypertension (stage I-II, stage I-II), which is established according to the classification of arterial hypertension (HTN) by stages, degrees and cardiovascular risk.

Accordingly, the indicators SBP within 140 - 159 mmHg, DBP 90 - 99 mmHg - HTN stage I;

SBP within 160 - 179 mmHg, DBP 100 - 109 mmHg - HTN stage II. Depending on the damage to target organs:

Stage I - objective signs of organic damage to target organs are absent; Stage II - there are objective signs of target organ damage without symptoms or dysfunction: LV hypertrophy (according to ECG, Echo-CG, MRI).

* reduced bone mineral density (BMD), which meets the criteria for osteopenia of the I-III degree, established by ultrasound densitometry: osteopenia of the I degree T-score from -1.0 to -1.5, II degree T-score from -1.5 to -2.0, III degree T-score from -2.0 to -2.5;
* patient's readiness for adequate cooperation in the process of clinical trials.

Exclusion Criteria:

* diagnosed congenital or acquired heart defects;
* established non-coronary myocardial diseases (myocarditis, cardiomyopathy);
* rhythm or conduction disorders with concomitant hemodynamic disorders (extrasystoles, paroxysmal tachycardias, atrial fibrillation/flutter, AV block 2 and 3 degrees);
* endocrine diseases, blood system diseases, systemic connective tissue diseases;
* diagnosed chronic obstructive pulmonary disease;
* impaired renal function (glomerular filtration rate according to the CKD-EPI formula less than 60 ml/min), liver.
* verified oncological diseases;
* abnormal uterine bleeding, endometriosis, pelvic inflammatory diseases;
* endometrial polyps and large uterine fibroids;
* inflammatory bowel diseases (IBD): Crohn's disease, nonspecific ulcerative colitis;
* hormone therapy;
* artificial early menopause;
* HIV/AIDS;
* alcohol or drug addiction;
* intolerance or allergic reaction to resveratrol, microcrystalline cellulose, grapes, red wine or blueberries;
* participation in other clinical trials

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 80 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
To measure the influence of trans-resveratrol on a development of chronic heart failure in early postmenopausal women period (1-4 years) with arterial hypertension and decreased bone mineral density | From enrollment to the end of treatment (3 month for each patient)
  * Percentage of patients in whom the use of 500 mg trans-resveratrol daily contributed to the normalization of laboratory and instrumental parameters;
  * Percentage of patients in whom the use of 500 mg trans-resveratrol daily contributed to the normalization of quality of life (according to the MENQOL and EuroQol-5D-3L questionnaires);
  * Percentage of patients in whom the use of 500 mg trans-resveratrol daily contributed to the reduction of risks of low-trauma fractures (according to the FRAX scale);
  * Percentage of patients in whom the use of 500 mg trans-resveratrol daily contributed to the reduction of cardiovascular risk (according to the SCORE2 algorithm and ST2 scale).
The safety of long-term using of trans-resveratrol in the amount of 500 mg per day | From enrollment to the end of treatment (3 month for each patient)
  The level of adverse events that does not exceed 5% of the sample size (N=50).

CONTACTS AND LOCATIONS:
Locations (1):
- Omnifarma LLC, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided